CLINICAL TRIAL: NCT04552561
Title: My MS Toolkit + Coaching: A Guided Web-based Symptom Self-Management Program for People With MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Anna Kratz, Associate Professor of Physical Medicine and Rehabilitation, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00184319
Record Dates: First submitted 2020-09-01; First posted 2020-09-17 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Multiple Sclerosis
Keywords: Self-management; Web-based program
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- My MS Toolkit (Experimental): 10 Participants asked to use My MS Toolkit and meet weekly with a study coach via telephone.
  Interventions: Behavioral: My MS Toolkit

INTERVENTIONS:
Behavioral: My MS Toolkit — My MS Toolkit, a web-based self-management intervention designed to help persons with Multiple Sclerosis self-manage fatigue, pain, and depressed mood.

SUMMARY:
My MS Toolkit is a web-based symptom self-management program for persons with multiple sclerosis (MS).

This study is evaluating various aspects of My MS Toolkit plus coaching and how it impacts symptom self-management in multiple sclerosis. The research team believe that the toolkit will be feasible, acceptable, and beneficial to participants.

DETAILED DESCRIPTION:
Study participants will be asked to use a newly developed web-based symptom self-management program, called the My MS Toolkit, for 8 weeks.

The My MS Toolkit includes 8 modules that describe symptom self-management strategies. Participants will explore the My MS Toolkit, following the prompts and guides built into the program, and meet with a study coach weekly for 15 to 30-minute telephone-delivered coaching sessions. Participants are encouraged to practice and apply the skills learned.

The study can be done from participants' homes using a reliable internet-connected device. No travel is required.

ELIGIBILITY:
Inclusion Criteria:

* Multiple Sclerosis
* Have access to a reliable, internet-connected device (e.g. computer, tablet). (Note: this study is conducted electronically and is not location dependent.)
* One or more of the following:

  1. Moderate/moderately severe depressive symptoms
  2. Chronic pain
  3. Presence of significant fatigue symptoms
* Read, speak and understand English.

Exclusion Criteria:

* Significant cognitive impairment
* Current psychotherapy for symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2021-01-18 (Actual); Study Completion 2021-01-18 (Actual)

PRIMARY OUTCOMES:
Acceptability/Feasibility of the the coached version of My MS Toolkit | Post-treatment, approximately week 8
  Assessed by the Participant Satisfaction Evaluation Survey. This survey is a 17 item scale with one free text item and 16 items with scores ranging from 1-4 (lowest to highest) with total scores ranging from 16-64. Higher scores indicate greater levels of acceptability.

SECONDARY OUTCOMES:
Impact of My MS Toolkit: Change in fatigue | Pre-treatment and Post-treatment, approximately week 8
  The Modified Fatigue Impact Scale will be used to assess fatigue. It is a self-report survey that contains 21 items. Each item is rated 0-4. Higher scores indicate a greater impact of fatigue on a person's activities.
Impact My MS Toolkit: Change in pain interference as measured by The Brief Pain Inventory Short Form | Pre-treatment and Post-treatment, approximately week 8
  The Brief Pain Inventory Short Form (BPI-SF) is a 9-item questionnaire (15 prompts) with two domains: pain severity and pain interference. The 7 pain interference items have values which range from 0 ("does not interfere") to 10 ("completely interferes"); items are averaged for a scale score range of 0-10, with higher scores indicating more pain interference.
Impact My MS Toolkit: Change in depressive symptoms as measured by the Patient Health Questionnaire depression scale | Pre-treatment and Post-treatment, approximately week 8
  The eight-item Patient Health Questionnaire depression scale (PHQ-8) is established as a valid diagnostic and severity measure for depressive disorders in large clinical studies. Scores range from 0 - 24 and a score of 10 or greater is consistent with at least moderate depressive symptoms.
Change in self-efficacy for managing symptoms as measured by the University of Washington Self-Efficacy Scale | Pre-treatment and Post-treatment, approximately week 8
  Changes measured by the University of Washington Self-Efficacy Scale (UW-SES), higher score indicates higher levels of self-efficacy (total score range: 6-30)
Participant perception of change | Post-treatment, approximately week 8
  Perception of change is assessed by the patient global impression of change questionnaire, which is 1 question and responses range from 1-7. Higher numbers indicate greater improvement in condition.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Kratz, Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No